CLINICAL TRIAL: NCT01801605
Title: Does Repetitive Transcranial Magnetic Stimulation (rTMS) Reduce Rectal Hypersensitivity in Patients With IBS ?
Brief Title: Repetitive Transcranial Magnetic Stimulation in Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 2007/053/HP; 2007-A00799-44
Record Dates: First submitted 2009-02-17; First posted 2013-03-01 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS - rectal hypersensitivity - rectal barostat - rTMS.
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- on (Active Comparator): active session
  Interventions: Procedure: rTMS
- off (Placebo Comparator): fictive session
  Interventions: Procedure: rTMS

INTERVENTIONS:
Procedure: rTMS — Active session with stimulation and placebo session with fictive stimulation
  Other Names: Active:A; Placebo:B

SUMMARY:
The purpose of this study is to evaluate the efficacy of Repetitive Transcranial Magnetic Stimulation (rTMS) on rectal hypersensitivity in patients with irritable bowel syndrome (IBS) in a prospective, randomized, double-blind study.

DETAILED DESCRIPTION:
IBS patients frequently demonstrate a rectal hypersensitivity which could participate to the abdominal pain. rTMS is an effective treatment of neurogenic chronic pain. The aim of the study is to evaluate the efficacy of rTMS on rectal hypersensitivity in patients with IBS in a prospective, randomized, double-blind study.

Patients and method: 20 patients with rectal hypersensitivity secondary to IBS will have one active session of rTMS located on the cortical area of the abdominal muscles during 5 consecutive days and one session of simulated rTMS during 5 over consecutive days corresponding to the placebo session. The order of the two session will be randomized. The efficacy of rTMS will be assessed by a rectal barostat to determine the pain or discomfort threshold and by a RIII reflex. The barostat and RIII reflex will be performed at the beginning and at the end of each session.

The investigators hope to demonstrate an improvement of the rectal hypersensitivity during the active stimulations compared to the placebo one.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old
* IBS defined by Rome III criteria
* Rectal hypersensitivity evaluated by barotat with a pain or inconfort volume less than 28 mmHg
* IBS for more than 3 months
* With an organic exploration for less than 6 months
* Without any knowledge concerning the rTMS

Exclusion Criteria:

* Pregnant women or women without any contraception
* Patients with pace-maker or other metallic implant
* Patients complaining of epilepsia or with past of epilepsia
* Patients with psychiatric disorders
* Patients treated by any drugs which could interfere with rTMS
* Patients having participate to another protocol within the month preceeding the inclusion
* Patients who could not stop the antalgic drugs within the week preceeding the onset of the study
* patients with a significant lesion on RMI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Pain or discomfort threshold volumes | final (up to 5 days)

SECONDARY OUTCOMES:
Amplitude of R3 reflex
Visual analogic scale
Symptoms diary
Quality of life scores

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie Leroi, phD, Principal Investigator — CHU Rouen
Locations (1):
- Physiology Unit-Rouen university Hospital, Rouen, France